CLINICAL TRIAL: NCT04903600
Title: Efficacy Assessment of Probiotics Fruit Vegetable Fiber Powder on Intestinal Health and Immune System Improvement in Human Trial
Brief Title: Efficacy Assessment of Probiotics Product on Intestinal Health and Immune System Improvement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chung Shan Medical University (Other)
Collaborators: TCI Co., Ltd. (Industry)
Responsible Party: Principal Investigator, Chin-Lin Hsu, Professor, Chung Shan Medical University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: CS2-21043
Record Dates: First submitted 2021-05-23; First posted 2021-05-26 (Actual); Last update posted 2021-09-14 (Actual); Status verified 2021-09

CONDITIONS: Healthy
MeSH Terms: interventions — Probiotics

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotics (Experimental): 32g probiotics fruit vegetable fiber powder product contained 1.12*10(11) CFU of probiotics for 12 weeks
  Interventions: Dietary Supplement: Probiotics fruit vegetable fiber powder product
- Placebo (Placebo Comparator): 32g placebo contained only maltodextrin (100%) for 12 weeks
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotics fruit vegetable fiber powder product — Eat 16 g for once, and twice a day
  Other Names: Probiotics
  Arms: Probiotics
Dietary Supplement: Placebo — Eat 16 g for once, and twice a day
  Arms: Placebo

SUMMARY:
The aim of this study is to investigate the effects of probiotics product (probiotics fruit vegetable fiber powder) on intestinal health and immune system improvement in adults

DETAILED DESCRIPTION:
This 12 weeks randomized, single-blind and placebo-controlled study will be conduct in fifty adults. Subjects will be recruited and assigned into two groups in a 1:1 ratio (placebo, n = 25; probiotics, n=25). During the 12 weeks intervention, the subjects should take 32 g powder of placebo or probiotics product (eat 16 g for once, and twice a day). The two powder supplied in an aluminum sachet, and all products were identical in taste. Subjects also should complete the assessment of anthropometric measurement, health conditions, food record, and sample collection (feces and blood) at week 0, 4, 8 and week 12.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion criteria include male or female participants to be aged 20-60 years old, who had colds more than four times in the past year or had gastric Infection by Helicobacter pylori or peptic ulcer, body mass index within a healthy range (18.5-27 kg/m2) and willing to commit throughout the experiment.

Exclusion Criteria:

* Exclusion criteria included cancer, chronic heart disease, use drugs which pharmacological effects may affect immunity, have systemic infections, use probiotics, prebiotics, fruit vegetable fiber supplementation, and lactose Intolerance or cow's milk allergic. Individuals who, in opinion of the investigator, seemed unlikely to complete the trial were also excluded.

Ages: 20 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-04-22 (Actual); Primary Completion 2021-09 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Change from baseline serum TNF-α at week 12 | Week0, Week12
  Compared the difference of serum cytokine TNF-α level between the week 12 and 0
Change from baseline serum IL-6 at week 12 | Week0, Week12
  Compared the difference of serum IL-6 level between the week 12 and 0
Change from baseline serum IL-10 at week 12 | Week0, Week12
  Compared the difference of serum IL-10 level between the week 12 and 0

CONTACTS AND LOCATIONS:
Overall Officials: Yu-Jou Chien, PhD Student, Principal Investigator — Chung Shan Medical University; Ying-Chi Chen, MS Student, Principal Investigator — Chung Shan Medical University
Locations (1):
- Chung Shan Medical University, Taichung, South, Taiwan